CLINICAL TRIAL: NCT04135365
Title: Identifying Modifiable Risk and Protective Factors for Neurocognitive Complications of Pediatric Type 1 Diabetes
Brief Title: Pediatric Type 1 Diabetes and Neurocognitive Complications Cohort Study
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sarah Jaser, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Other Study IDs: T1DCohortStudy; 1U34DK123895-01 (NIH)
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric T1D: A sample of 20 children with Type 1 Diabetes and their caregivers will be asked to stay after their diabetes clinic appointment to complete enrollment, or they may choose to come back for a study visit. Trained study staff will describe the study in detail to interested families. They will be encouraged to ask questions before giving consent. After obtaining informed consent/assent, children and caregivers will schedule time for a neurocognitive assessment and neuroimaging assessment. Children and caregivers will complete assessments again approximately 12 months later.
  Interventions: Behavioral: neurocognitive assessment; Behavioral: neuroimaging assessment
- Comparison: Children with no known chronic medical conditions or intellectual disability will undergo the same procedure listed for the Pediatric T1D group
  Interventions: Behavioral: neurocognitive assessment; Behavioral: neuroimaging assessment

INTERVENTIONS:
Behavioral: neurocognitive assessment — Observational study therefore there are no interventions
Behavioral: neuroimaging assessment — Observational study therefore there are no interventions

SUMMARY:
The proposed project will assess hypothesized risk factors (age of onset, Diabetic ketoacidosis (DKA) at presentation and glycemic control), as well as potentially modifiable protective factors (child sleep quality, caregiver distress, and use of diabetes devices). In addition, the study will optimize imaging protocols and processing tools to allow for harmonization of neuroimaging data across sites and scanners for the most robust analysis.

DETAILED DESCRIPTION:
The onset of type 1 diabetes (T1D) in childhood results in clinically significant deficits in neurocognitive functioning that manifest in adulthood. These deficits have implications for adaptive functioning and diabetes management. Studies of neurocognitive function and brain development in T1D suggest that factors such as age of onset, diabetic ketoacidosis (DKA) at time of onset, and exposure to chronic hyperglycemia or severe hypoglycemia may increase risk or severity of these deficits, but findings are mixed. The majority of previous studies were limited by the use of adult or older adolescent samples, cross-sectional designs or short duration of follow-up, lack of racial and ethnic diversity, and small sample sizes. Age-related changes in neurocognitive function and vascular complications associated with T1D in adults make isolating mechanisms more complex. The knowledge gaps are critical because individuals with T1D may live for decades with reduced neurocognitive function. Building on previous work, it is hypothesized that several risk and protective factors for neurocognitive deficits will be evident in youth with T1D. First, sleep is a critical and potentially modifiable risk or protective factor for youth. Prior work has shown that the majority of school-age children do not obtain sufficient sleep (67%), and that sleep disturbances are related to poor glycemic control and risk for DKA, both of which have been posited to increase risk for neurocognitive deficits. Second, caregiver distress (i.e., symptoms of anxiety and depression) is a significant risk factor for child wellbeing, as exposure to maternal depressive symptoms increases children's risk for cognitive deficits and abnormal white matter diffusivity. Third, improved glycemic control via use of continuous glucose monitors and hybrid closed-loop insulin delivery systems, are potential protective factors for youth with T1D, as these devices decrease glycemic variability and limit time spent in hypoglycemia and hyperglycemia. Thus, a prospective longitudinal cohort study of young children with T1D is needed to identify modifiable risk and protective factors for neurocognitive complications. If specific risk or protective factors for adverse or optimal neurocognitive outcomes are defined, treatment protocols could be developed to limit neurocognitive complications associated with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric T1D sample: Children will be eligible if they meet the following inclusion/exclusion criteria:

  1. are between 6 -11 years of age
  2. have no history of afebrile seizure (not related to hypoglycemia) or sleep disorders other than insufficient sleep or insomnia
  3. no contraindications to high quality MRI of the brain (no metal implants or braces)
  4. no premature birth (<34 weeks) or low birth weight (<2,000g).

Comparison sample: Children will be eligible if they meet the following inclusion/exclusion criteria:

1. no known chronic medical conditions or intellectual disability
2. no known history of concussion or traumatic brain injury
3. no history of afebrile seizure; (4) no braces or metal implants

(5) no premature birth (<34 weeks) or low birth weight (<2,000g).

Parents or primary caregivers of all children will be eligible if they:

1. live with the child
2. read/speak English to allow use of validated parental questionnaires. The parent who is the primary caregiver of the child will be invited to participate.

Exclusion Criteria:

* N/A

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The Children's Diabetes Program (CDP) at Vanderbilt University Medical Center in collaboration with strong multidisciplinary research collaborators is well poised to answer these questions with considerable local expertise in behavioral research in children with T1D, neurocognitive testing in youth with T1D, pediatric neurology and neuroimaging, and data science. Further, we bring unique expertise in sleep in youth with T1D, caregiver distress, and use of novel measurement tools. Finally, the CDP follows over 2,800 children with diabetes, 85% of whom have T1D, and there are about 250 new-onset cases of T1D annually.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Cognitive Function: Full-scale IQ | 12 months
  To assess cognitive differences in full-scale IQ using the Wechsler Intelligence Scale for Children, fifth edition (WISC V) in children with T1D vs. comparison children. The Full-Scale IQ is an estimate of overall intellectual ability. The WISC-V takes approximate 48 minutes to administer. The FSQI uses a standard score metric with a mean of 100 and an Standard Deviation of 15.
Cognitive Function: Executive Function | 12 monnths
  To assess cognitive differences in executive function using the The NIH Toolbox Executive Function Tests in children with T1D vs. comparison children.
  1) NIH Flanker Inhibitory Control and Attention Test will be used to assess children's ability to inhibit visual attention. Average administration time is 4 minutes. A scoring algorithm integrates accuracy, a suitable measure in early childhood, yielding scores from 0 to 10.
Cognitive Function: Behavior Rating Inventory of Executive Function, Second Edition | 12 months
  Parent report of child's executive function, has been validated for use in children ages 5-18 years. Scaled T-scores are based on normative data for age and sex. The BRIEF2 consists of 63 items, and it yields a Global Executive Composite score, as well as a Behavior Regulation Index, Emotional Regulation Index, and Cognitive Regulation Index

SECONDARY OUTCOMES:
Imaging | 12 months
  Differences in brain volume and white matter microstructure in children with T1D vs comparison children.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah S Jaser, PhD, Principal Investigator — Vanderbilt University Medical Center; Lori Jordan, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All of our de-identified data will be stored in REDCap. Other researchers will be required to register with REDCap and agree to conditions listed in REDCap governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. REDCap offers a mechanism to allow third parties to track de-identified data downloads and datasets to users with specific access granted. Data may be downloaded in several file formats including STAT, SAS, R, and Excel. The ability to share MRI data will be limited by file size, costs and time to transmit imaging. Our study imaging scientists will create methods for secure sharing of imaging data. If source imaging data is requested, any costs to share these data would need to be arranged by the requesting investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available to external investigators within five years after study completion and after the publication of study results.
Access Criteria: Investigators are required to submit a proposal requesting: Investigator's name and affiliation; Hypothesis to be tested or investigation to be conducted; Background and relevant literature; Subjects eligible for inclusion in the analysis and dataset; List of variables of interest; Substantially detailed analysis plan; List of potential co-authors and collaborators. The proposal must be submitted to the Co-PI and will be reviewed by KSP. The PI and statistician will send a confidentiality agreement stipulating that the data file is to be used only for the purpose described in the proposal and that the requesting investigator must retain control over the file at all times. The requesting investigator is further obligated to supply quarterly progress reports on their analysis/investigation and to supply draft manuscripts. Prior to the release of the file, the contact PI and statistician will personally review the file and certify the level of de-identification.